CLINICAL TRIAL: NCT06509607
Title: Effects of Lower Limb Concentric Versus Eccentric Dynamic Resistance Training on Agility and Speed in Badminton Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0486 Umar
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Sports Physical Therapy
Keywords: Agility; Badminton; Concentric Training; Dynamic resistance training; Speed; Eccentric training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 32 participants will be in experimental group A and will perform concentric lower limb training program including squats, lunges and leg extension exercises.
  Interventions: Other: Concentric Lower Limb Training Program
- Group B (Experimental): 32 participants will be in experimental group B and will perform eccentric lower limb training program including wall sit, sitting straddle single leg and full squat exercises.
  Interventions: Other: Eccentric Lower Limb Training Program

INTERVENTIONS:
Other: Concentric Lower Limb Training Program — A specially designed 30-minute concentric lower limb training program (squats, lunges and leg extensions) conducted by the researchers, before a 90-minute ordinary badminton training session conducted by the coach, 2 days per week for 8 weeks.
  Arms: Group A
Other: Eccentric Lower Limb Training Program — A specially designed 30-minute eccentric lower limb training program (wall sit, sitting straddle single leg and full squat) conducted by the researchers, before a 90-minute ordinary badminton training session conducted by the same coach, 2 days per week for 6 weeks.
  Arms: Group B

SUMMARY:
With an average heart rate (HR) of more than 90% of the player's maximal HR, football is extremely taxing. The sporadic movements that occur throughout a game place a strain on the anaerobic and aerobic systems, accounting for roughly 30% of the latter's workload and 60% of the former. The capacity to shift directions and accelerate or decelerate on the court in order to make accurate shots and perform better is what determines footwork performance. Plyometric Training is a favored training technique for raising COD performance since it has a reputation for being a simple, quick, and efficient method of training. The core practice of combining resistance conditioning exercises with a dynamic warm-up can improve power output in badminton and create a post-activation performance enhancement (PAPE) impact. According to random sampling and sample size calculated by open epi tool, a total of 68 badminton players will be obtained from the badminton club of a Crescent sports club and Al-Fatah Sports Complex, Faisalabad. They will be divided into group A and group B according to the form of random sampling. Baseline markers for agility and speed will be taken before the start of the training and after the completion of training program. Group A will be engaged in a specially designed 30-minute concentric lower limb training program (squats, lunges and leg extensions) conducted by the researchers, before a 90-minute ordinary badminton training session conducted by the coach, 2 days per week for 8 weeks. Group B will be engaged in a specially designed 30-minute eccentric lower limb training program (wall sit, sitting straddle single leg and full squat) conducted by the researchers, before a 90-minute ordinary badminton training session conducted by the same coach, 2 days per week for 8 weeks.

DETAILED DESCRIPTION:
The aim of the study is to find out the effects of concentric and eccentric dynamic resistance training on agility and speed in badminton players

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 (12)
* Both male & female players
* Healthy players/no injuries (8)
* No severe injuries during the last six months (16)
* Player with minimum 1-year experience of badminton (17)

Exclusion Criteria:

* Serious musculoskeletal injuries/disorders(8)
* Participants who will be unable to complete concentric/eccentric dynamic resistance training
* Who will be unwilling to complete six-weeks of training and tests

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Lateral Change of Direction Test | 8 weeks
  To perform the test, the athlete warms up for 10 minutes The assistant places three cones 5 metres apart on a straight line The athlete stands by the middle cone (B), facing the assistant The assistant gives the command "GO" and points in a starting direction, right or left, and starts the stopwatch The athlete moves to and touches the first cone, returns past the middle cone to the far cone and touches it and then returns to and touches the middle cone The assistant stops the stopwatch when the athlete touches the middle cone and records the time The test is conducted four times - two in each starting direction (left & right) The fastest time in each direction is used for accessing the athlete's performance
60 Metre Speed Test | 8 weeks
  This test requires the athlete to sprint as fast as possible over 60 metres
  The athlete warms up for 10 minutes The assistant marks out a 60-metre straight section on the track with cones The assistant gives the command "GO" and starts the stopwatch The athlete sprints as fast as possible over the 60 metres The assistant stops the stopwatch as the athlete's torso crosses the finishing line and records the time The test is conducted three times The assistant uses the fastest recorded time to assess the athlete's performance

CONTACTS AND LOCATIONS:
Overall Officials: Muzna Munir, Ppdpt, Principal Investigator — Riphah International University
Locations (1):
- Crescent Sports Complex, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabello-Manrique D, Lorente JA, Padial-Ruz R, Puga-Gonzalez E. Play Badminton Forever: A Systematic Review of Health Benefits. Int J Environ Res Public Health. 2022 Jul 26;19(15):9077. doi: 10.3390/ijerph19159077. PMID 35897446
- [Background] Edel A, Weis JL, Ferrauti A, Wiewelhove T. Training drills in high performance badminton-effects of interval duration on internal and external loads. Front Physiol. 2023 Jun 30;14:1189688. doi: 10.3389/fphys.2023.1189688. eCollection 2023. PMID 37457032
- [Background] Asadi A, Arazi H, Young WB, Saez de Villarreal E. The Effects of Plyometric Training on Change-of-Direction Ability: A Meta-Analysis. Int J Sports Physiol Perform. 2016 Jul;11(5):563-73. doi: 10.1123/ijspp.2015-0694. Epub 2016 May 3. PMID 27139591
- [Background] Santoro E, Tessitore A, Liu C, Chen CH, Khemtong C, Mandorino M, Lee YH, Condello G. The Biomechanical Characterization of the Turning Phase during a 180 degrees Change of Direction. Int J Environ Res Public Health. 2021 May 21;18(11):5519. doi: 10.3390/ijerph18115519. PMID 34063934
- [Background] Chua MT, Chow KM, Lum D, Tay AWH, Goh WX, Ihsan M, Aziz AR. Effectiveness of On-Court Resistive Warm-Ups on Change of Direction Speed and Smash Velocity during a Simulated Badminton Match Play in Well-Trained Players. J Funct Morphol Kinesiol. 2021 Sep 27;6(4):81. doi: 10.3390/jfmk6040081. PMID 34698234
- [Background] Condello G, Minganti C, Lupo C, Benvenuti C, Pacini D, Tessitore A. Evaluation of change-of-direction movements in young rugby players. Int J Sports Physiol Perform. 2013 Jan;8(1):52-6. doi: 10.1123/ijspp.8.1.52. Epub 2012 Jul 31. PMID 22869638
- [Background] Malwanage KT, Senadheera VV, Dassanayake TL. Effect of balance training on footwork performance in badminton: An interventional study. PLoS One. 2022 Nov 17;17(11):e0277775. doi: 10.1371/journal.pone.0277775. eCollection 2022. PMID 36395192
- [Background] Phomsoupha M, Laffaye G. The science of badminton: game characteristics, anthropometry, physiology, visual fitness and biomechanics. Sports Med. 2015 Apr;45(4):473-95. doi: 10.1007/s40279-014-0287-2. PMID 25549780
- [Background] Yeung WV, Bishop C, Turner AN, Maloney SJ. Does a Loaded Warm-Up Influence Jump Asymmetry and Badminton-Specific Change of Direction Performance? Int J Sports Physiol Perform. 2021 Apr 1;16(4):578-584. doi: 10.1123/ijspp.2020-0313. Epub 2021 Jan 31. PMID 33524952
- [Background] Sonoda T, Tashiro Y, Suzuki Y, Kajiwara Y, Zeidan H, Yokota Y, Kawagoe M, Nakayama Y, Bito T, Shimoura K, Tatsumi M, Nakai K, Nishida Y, Yoshimi S, Aoyama T. Relationship between agility and lower limb muscle strength, targeting university badminton players. J Phys Ther Sci. 2018 Feb;30(2):320-323. doi: 10.1589/jpts.30.320. Epub 2018 Feb 28. PMID 29545704